CLINICAL TRIAL: NCT04624295
Title: Early Antiplatelet Therapy After Hemorrhagic Infarction in Acute Ischemic Stroke Treated With Intravenous Thrombolysis in China (HITs)：a Randomized Clinical Trial
Brief Title: Early Antiplatelet Therapy After Hemorrhagic Infarction in Acute Ischemic Stroke Treated With Intravenous Thrombolysis (HITs)
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: Shaoxing People's Hospital (Other); Affiliated Hospital of Jiaxing University (Other); Huzhou Central Hospital (Other); The Second Affiliated Hospital of Jiaxing University (Other); Jinhua Central Hospital (Other); Taizhou Hospital (Other); Ningbo Medical Center Lihuili Hospital (Other Government); Ningbo No.2 Hospital (Other); Lishui Country People's Hospital (Other); Wenzhou Central Hospital (Other); The Fourth Affiliated Hospital of Zhejiang University School of Medicine (Other); Shenzhen Second People's Hospital (Other); The Affiliated Hospital of Xuzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HITs
Record Dates: First submitted 2020-10-29; First posted 2020-11-10 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-05

CONDITIONS: Antiplatelet Therapy; Hemorrhagic Infarction
Keywords: acute ischemic stroke; intravenous thrombolysis; Hemorrhagic Infarction; antiplatelet therapy
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Early Antiplatelet Therapy (Active Comparator)
  Interventions: Drug: Early aspirin Therapy
- Non-Early Antiplatelet Therapy (Placebo Comparator)
  Interventions: Drug: Non-Early aspirin Therapy

INTERVENTIONS:
Drug: Early aspirin Therapy — Early Antiplatelet Therapy is administered within 24 to 48 hours after stroke onset and the dose is determined by the clinician. Aspirin was chosen for antiplatelet therapy.
  Arms: Early Antiplatelet Therapy
Drug: Non-Early aspirin Therapy — Antiplatelet therapy will be delayed to beyond 48 hours after stroke onset and may not be initiated until hemorrhagic Infarction has been confirmed absorbed.
  Arms: Non-Early Antiplatelet Therapy

SUMMARY:
Previous study showed that the proportions of hemorrhagic Infarction after intravenous thrombolysis were 24.2% and 32.5% in the control group and the alteplase group, and most of them were asymptomatic. Hemorrhagic Infarction was a part of the natural progression after acute ischemic stroke. Previous study have shown no significant relationship between hemorrhagic Infarction and poor outcome in acute ischemic stroke (AIS) patients. In this study, a randomized controlled trial will be conducted to explore the efficacy and safety of early antiplatelet therapy after hemorrhagic infarction in acute ischemic stroke treated with intravenous thrombolysis.

ELIGIBILITY:
Inclusion Criteria:

1. Acute ischemic patients receiving intravenous thrombolysis within 24 hours upon stroke onset
2. Be confirmed as Hemorrhagic Infarction at 24 to 36 hours after intravenous thrombolysis by computerized tomography
3. The patient or family member signed an informed consent

Exclusion Criteria:

1. Early use of anticoagulant drugs within 1 week after intravenous thrombolysis;
2. Tirofiban was used after receiving endovascular treatment;
3. Intraoperative stent placement after receiving endovascular treatment;
4. Subarachnoid hemorrhage or ventricular hemorrhage;
5. There are contraindications for aspirin use;

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 294 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
The proportion of patients with modified Rankin scale (mRS) ≤2 | 90 days
  The proportion of patients with modified Rankin scale (mRS) ≤2 at 90 days, on which scores range from 0 (no neurologic deficit) to 6 (death)].

SECONDARY OUTCOMES:
Hemorrhage enlargement after intravenous thrombolysis | 7 days
  Hemorrhage enlargement after intravenous thrombolysis at 7 days
Hemorrhage reduction after intravenous thrombolysis | 7 days
  Hemorrhage reduction after intravenous thrombolysis at 7 days
the progress of National Institute of Health Stroke Scale (NIHSS) scores | 7 days
  the progress of National Institute of Health Stroke Scale (NIHSS) scores at 7 days, on which scores range from 0 (no neurologic deficit) to 42 (severe)]
the distribution of modified Rankin scale (mRS) | 90 days
  the distribution of modified Rankin scale (mRS) at 90 days, on which scores range from 0 (no neurologic deficit) to 6 (death)]
Recurrence rate of acute ischemic stroke | 90 days
  Recurrence rate of acute ischemic stroke at 90 days
Recurrence rate of cerebrovascular disease | 90 days
  Recurrence rate of cerebrovascular disease at 90 days
Recurrence rate of acute ischemic stroke | 1 year
  Recurrence rate of acute ischemic stroke at 1 years
Recurrence rate of cerebrovascular disease | 1 year
  Recurrence rate of cerebrovascular disease at 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Min Lou, PhD, Study Director — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (1):
- the second affiliated hospital of Zhejiang University, Hangzhou, China

IPD SHARING:
Plan to Share IPD: No